CLINICAL TRIAL: NCT01880112
Title: Serum and Tissue Cefazolin Concentrations in Normal Weight Patients Undergoing Cesarean Delivery Receiving Two Differing Doses of Pre-operative Cefazolin.
Brief Title: Serum and Tissue Cefazolin Concentrations in Normal Weight Patients Undergoing Cesarean Delivery.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: There is no longer need for this study.
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Michael Stitely, Adjunct Associate Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H-23256
Record Dates: First submitted 2011-06-29; First posted 2013-06-18 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Infection; Cesarean Delivery; Antibiotic Prophylaxis
Keywords: Infection; Cesarean delivery; Antibiotic prophylaxis; Cefazolin dosing
MeSH Terms: conditions — Infections | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4 gram dose (Experimental): Pre-operative prophylactic dose of 4 grams of cefazolin
  Interventions: Drug: Cefazolin
- 2 gram dose (Active Comparator): Pre-operative prophylactic dose of 2 grams of cefazolin
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — Cefazolin will be administered as pre-operative prophylaxis in normal weight patients undergoing Cesarean delivery. Tissue and serum levels will be measured at the time of the incision and when the incision is closed.
  Other Names: Ancef

SUMMARY:
Patients undergoing Cesarean delivery (C-Section) with a body mass index of 30 or less will be given either 2 grams or 4 grams of an antibiotic before surgery. The antibiotic is intended to prevent infection from the surgery. It is unknown what the best dose for the usual medicine used for this purpose (an antibiotic medicine called cefazolin). Samples of the tissue just under the skin will be biopsied at the time the incision is made and at the time the cut is stitched or stapled closed. A sample of the muscle of the womb will be taken as the womb is stitched closed after the delivery. Blood tests will be done at the start and end of surgery to test the antibiotic level. A blood sample will be taken from the umbilical cord after the baby has been delivered and the umbilical cord has been cut. The umbilical cord blood sample will be tested for the antibiotic level. These tests will be used to find out if the usual dose of medicine is enough or if more medicine is needed to prevent infection in normal weight women undergoing c-sections.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above
2. Body mass index (BMI) of 30 or less, as calculated from the height and weight at the first prenatal visit
3. Undergoing cesarean delivery

Exclusion Criteria:

1. BMI greater than 30.
2. Not undergoing Cesarean delivery.
3. Age less than 18 years.
4. Pre-existing infection.
5. Allergy to cephalosporin medications or a history of an anaphylactic reaction to penicillin.
6. Cesarean delivery being performed under emergent circumstances

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Cefazolin drug level. | Tissue and blood samples will be drawn during the surgical case only. Duration expected to be less than 120 minutes.
  Measurement of the serum and tissue level of cefazolin.

CONTACTS AND LOCATIONS:
Overall Officials: William H Holls, MD, Principal Investigator — West Virginia University; Michael L Stitely, MD, Study Chair — West Virginia University
Locations (1):
- West Virginia University Hospital, Morgantown, West Virginia, United States